CLINICAL TRIAL: NCT05100082
Title: Special Drug Use Surveillance for Cabometyx Tablets "Hepatocellular Carcinoma"
Brief Title: Survey of Cabozantinib Tablets Used To Treat People With Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Cabozantinib-5002; jRCT2031210403 (Registry Identifier: jRCT)
Record Dates: First submitted 2021-10-28; First posted 2021-10-29 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Hepatocellular Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — cabozantinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cabozantinib 60 mg: Cabozantinib 60 milligrams (mg) tablet, orally, once daily for up to 12 months. Participants received interventions as part of routine medical care.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — Cabozantinib tablets
  Other Names: Cabometyx tablets

SUMMARY:
This study is a survey in Japan of Cabozantinib tablets used to treat Japanese people with a type of liver cancer called hepatocellular carcinoma. The study sponsor will not be involved in how the participants are treated but will provide instructions on how the clinics will record what happens during the study.

The main aim of the study is to check for side effects from Cabozantinib. During the study, participants with hepatocellular carcinoma will take Cabozantinib tablets according to their clinic's standard practice. The study doctors will check for side effects from Cabozantinib for 12 months.

ELIGIBILITY:
Inclusion Criteria:

Participants with unresectable hepatocellular carcinoma that has progressed after cancer chemotherapy (Regardless of previous treatment history)

Exclusion Criteria:

Participants who has a history of hypersensitivity to any component of cabozantinib.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with unrespectable hepatocellular carcinoma that has progressed after cancer chemotherapy in part of routine medical care.
Sampling Method: Probability Sample
Enrollment: 263 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events Related to Hepatic Failure, Hepatic Dysfunction, and Pancreatitis | Up to 12 months
  An adverse event (AE) is any untoward or undesirable medical occurrence in a participant linked in time with the use of a pharmaceutical/ medicinal product. They are not limited to the events with clear causal relationship with treatment with concerned drug. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
Number of Participants with Serious Adverse Events | Up to 12 months
  A serious AE is any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability / incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the above mentioned criteria.
Number of Participants with Adverse Events Leading to Permanent Treatment Discontinuation with Cabozantinib Tablets | Up to 12 months
Number of Participants with Grade 3 or higher Adverse Events | Up to 12 months
  Severity grade is defined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.

SECONDARY OUTCOMES:
Percentage of Participants Who Achieve or Maintain Any Best Response Category Assessed by Response Evaluation Criteria in Solid Tumors (RECIST 1.1) | Up to 12 months
  Best response will be assessed with reference to the excerpts from Response Evaluation Criteria in Solid Tumors (RECIST 1.1). Best response is defined as the level of best response in assessment with complete response (CR), partial response (PR), progressive disease (PD), stable disease (SD) and not evaluable (NE) during the observational period.
Percentage of Participants Who Achieve or Maintain Any Best Response Category Assessed by Modified Response Evaluation Criteria in Solid Tumors (Modified RECIST) | Up to 12 months
  Best response will be assessed with reference to the excerpts from Modified Response Evaluation Criteria in Solid Tumors (Modified RECIST). Best response is defined as the level of best response in assessment with CR, PR, PD, SD and NE during the observational period.
Disease Control Rate (DCR) | Up to 12 months
  DCR was defined as the percentage of participants whose best overall response is CR, PR or SD, per RECIST 1.1. CR was defined as disappearance of all target lesions; PR was defined as at least a 30% decrease in the sum of diameter (SoD) of target lesions, taking as a reference the baseline SoD. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Overall Survival (OS) | Up to 12 months
  OS is defined as time from the first day of study drug administration to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda Selected Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/6181fed7eb0e19002afd69f3